CLINICAL TRIAL: NCT02231762
Title: Phase II, Multicentre, Open Label Study to Evaluate the Efficacy of the Combination of Lanreotide Autogel 120mg and Temozolomide in Patients With Progressive Gastro-entero-pancreatic Neuroendocrine Tumours (GEP-NET) G1/G2 - A Pilot-Study
Brief Title: Combination of Lanreotide Autogel 120mg and Temozolomide in Progressive GEP-NET
Acronym: SONNET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-94-52030-268; 2013-001697-17 (EudraCT Number)
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-02

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lanreotide Autogel 120mg & Temozolomide (Experimental): Combination phase for first 6 months: Lanreotide Autogel 120 mg and Temozolomide.
  Followed by either 6 months Lanreotide Autogel 120 mg maintenance or 6 months of no treatment.
  Interventions: Drug: Lanreotide Autogel 120 mg; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Lanreotide Autogel 120 mg — Lanreotide Autogel 120 mg subcutaneous (s.c) - injection, every 28 days (+/-2 days).
Drug: Temozolomide (TMZ) — Temozolomide capsule (variable dose). 150 mg/m2 per day for 5 days in the first month. 200 mg/m2 per day for 5 days in months 2, 3, 4, 5 and 6.

SUMMARY:
The purpose of the study is to evaluate the efficacy and tolerability of the combination of Lanreotide Autogel 120 mg and Temozolomide in patients with progressive gastro-entero-pancreatic neuroendocrine tumours (GEP-NET) graded as G1 or G2 (G1/G2). All progressive tumours classified according to Response Evaluation Criteria In Solid Tumours (RECIST, 1.1).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study related procedures
* Inoperable, Gastro-Entero-Pancreatic-Neuroendocrine Tumour G1 or G2 (Proliferation Index, Ki67-Index: 0 to ≤20%) confirmed by pathological/histological assessment
* Progressive disease within 12 months before inclusion (RECIST 1.1: increase of >20% tumour load; by Computer Tomography (CT) or Magnetic Resonance Imaging (MRI)
* Measurable disease according to RECIST 1.1.
* Metastatic disease confirmed by CT/MRI.
* Functioning or non-functioning NET (G1, G2).
* Positive Octreo-Scan (≥ Grade 2 Krenning scale) or positive DOTA (1,4,7,10-tetraazacyclododecane-1,4,7,10-tetraacetic acid)-TATE (Tyr3-Thre8-Octreotide or DOTA-Tyr3-octreotate)/TOC (Tyr3-octreotide) -PET (Positron-Emission-Tomography) -CT within 12 months prior to screening

Exclusion Criteria:

* Has the diagnosis of Insulinoma
* Has a diagnosis of a multiple endocrine neoplasia (MEN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (10):
- Vienna General Hospital, Vienna, Austria
- Germany (9):
  - Zentralklinik Bad Berka, Bad Berka
  - Charité University Hospital, Berlin
  - University Hospital Essen, Essen
  - ENDOC Hamburg, Hamburg
  - Oncological Center Leer, Leer
  - University Hospital Mainz, Mainz
  - University Hospital Mannheim, Mannheim
  - University Hospital Marburg, Marburg
  - University Hospital Munich, Munich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 57 subjects entered a combination phase and received lanreotide ATG 120 mg plus temozolomide for 6 months. A 6 month maintenance phase then followed where subjects received either lanreotide ATG 120 mg or no treatment, dependent upon whether they had functioning or non-functioning NET, clinical benefit and allocation following randomisation.
Pre-assignment Details: Overall, 64 subjects were screened, 7 were screening failures of which 5 subjects did not meet the entry criteria. 57 subjects were assigned to receive treatment in the baseline population.
Groups:
- Combination Phase: All subjects received lanreotide ATG 120 mg plus temozolomide in combination for 6 months.
  Subjects received 1 injection of lanreotide ATG 120 mg and temozolomide capsules for 5 consecutive days, in a 28 day treatment cycle. The temozolomide dose was adapted to the subject body surface area (BSA) and the dose in the 1st treatment cycle was 150 mg/metres squared (m^2) per day. Depending on the safety laboratory values, the temozolomide dose was increased to 200 mg/m^2 per day from cycle 2 to cycle 6.
- Maintenance Phase - Functioning NET, Lanreotide: In case of clinical benefit, defined as either complete response (CR), partial response (PR) or stable disease (SD) after the first 6 months combination phase, all subjects with functioning (serotonin producing) NET continued to receive lanreotide ATG 120 mg for another 6 months. This maintenance phase started with visit 8, week 24.
- Maintenance Phase - Non-functioning NET, Lanreotide: Following completion of the 6-month combination phase, all subjects with non-functioning NET and clinical benefit were randomised to continue to receive lanreotide ATG 120 mg for another 6 months. This maintenance phase started with visit 8, week 24.
- Maintenance Phase - Non-functioning NET, No Treatment: Following completion of the 6-month combination phase, all subjects with non-functioning NET and clinical benefit were randomised to receive no treatment for 6 months. This maintenance phase started with visit 8, week 24.
Period: Combination Phase
Arm/Group | Combination Phase | Maintenance Phase - Functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, No Treatment
Started | 57 | 0 (This arm was not included in period 1 (combination phase).) | 0 (This arm was not included in period 1 (combination phase).) | 0 (This arm was not included in period 1 (combination phase).)
Completed | 37 | 0 | 0 | 0
Not Completed | 20 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Disease Progression | 6 | 0 | 0 | 0
Not completed — Did not meet inclusion criteria | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | Combination Phase | Maintenance Phase - Functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, No Treatment
Started | 0 (This arm was not included in period 2 (maintenance phase).) | 11 (The 37 subjects completing period 1 were split between the 3 arms in period 2.) | 14 (The 37 subjects completing period 1 were split between the 3 arms in period 2.) | 12 (The 37 subjects completing period 1 were split between the 3 arms in period 2.)
Completed | 0 | 8 | 9 | 7
Not Completed | 0 | 3 | 5 | 5
Not completed — Disease progression | 0 | 3 | 4 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Combination Phase
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native. | 0
  Asian. | 0
  Black or African American | 0
  Hispanic or Latino | 0
  Native Hawaiian or Other Pacific Islander. | 0
  White | 57

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR) After 6 Months
Description: All tumour assessments were performed using the Response Evaluation Criteria In Solid Tumours (RECIST) criteria (1.1). Computer Tomography (CT-scan) or Magnetic Resonance Imaging (MRI) could be used for as method of tumour measurement and the same method of tumour measurement was used throughout the study for each subject. CT scans/MRI were performed at screening or baseline visit then at weeks 12, 24 and at early withdrawal or at anytime during the study in the case of any clinical or biological signs of tumour progression.
  The DCR was defined as the proportion of subjects with a response of CR, PR or SD after 6 months of combination treatment and was described in the ITT population along with its 95% Confidence Interval (CI) and was compared to 45% with an exact binomial proportion test. The Last Observation Carried Forward (LOCF) method was used to replace missing assessments at the end of the combination phase.
Time Frame: 6 months
Population: The ITT population is all subjects that had at least one baseline and at least one post baseline assessment of the primary efficacy parameter.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Combination Phase
Number analyzed (Participants) | 49
percentage of subjects | 73.5 [58.9 to 85.1]

2. Secondary Outcome: DCR After 12 Months
Description: All tumour assessments were performed using the RECIST criteria (1.1). CT-scan or MRI could be used for as method of tumour measurement and the same method of tumour measurement was used throughout the study for each subject. CT scans/MRI were performed at screening or baseline visit then at baseline, weeks 12, 24, 36, 48 (end of study) and at study withdrawal or at anytime during the study in the case of any clinical or biological signs of tumour progression.
  The DCR was defined as the proportion of subjects with a response of CR, PR or SD after 6 months combination treatment followed by either 6 months of lanreotide ATG 120 mg maintenance treatment or no treatment. The DCR was described in the ITT population along with its 95% CI and was compared to 45% with an exact binomial proportion test. The LOCF method was used to replace missing assessments at the end of the maintenance phase.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Maintenance Phase - Non-functioning NET, Lanreotide: After the first 6 months combination phase, subjects with non-functioning NET and clinical benefit were randomised to continue to receive lanreotide ATG 120 mg for another 6 months. This maintenance phase started with visit 8, week 24.
- Maintenance Phase - Non-functioning NET, No Treatment: After the first 6 months combination phase, subjects with non-functioning NET and clinical benefit were randomised to receive no treatment for 6 months. This maintenance phase started with visit 8, week 24.
Arm/Group | Maintenance Phase - Functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, No Treatment
Number analyzed (Participants) | 11 | 14 | 12
percentage of subjects | 54.5 [23.4 to 83.3] | 71.4 [41.9 to 91.6] | 41.7 [15.2 to 72.3]

3. Secondary Outcome: Progression-Free Survival (PFS) Within 12 Months
Description: PFS was defined as the time from the date of treatment start to the date of the first documented disease progression or death due to any cause within the first 12 months of treatment. If a subject had not progressed or died after 12 months of treatment or when any further anti-neoplastic therapy was received, PFS was censored at the time of the last tumour assessment before the analysis cut-off date or the anti-neoplastic therapy date.
  A Kaplan-Meier estimate of the PFS was calculated to determine the number of subjects at risk. Median PFS time (50% of subjects who would not progress or die) of the ITT population is presented along with 95 % CI.
Time Frame: 12 months
Population: The ITT population is all treated subjects that had at least one baseline and at least one post baseline assessment of the primary efficacy parameter.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Intention-to-treat (ITT) Population: All treated subjects having at least one baseline and at least one post baseline assessment of the primary efficacy parameter.
Arm/Group | Intention-to-treat (ITT) Population
Number analyzed (Participants) | 49
months | 11.1 [8.3 to NA] — Upper limit of the 95 % CI could not be determined as too few survival events for complete data estimation were observed during the 12 month study duration.

4. Secondary Outcome: Time To Response (TtR) Within 12 Months
Description: TtR was defined as the time from the date of treatment start to the date of the first documented objective response (CR or PR) within the first 12 months of treatment (combination and maintenance phases). A Kaplan Meier estimate of the TtR survival function was constructed.
  The Kaplan-Meier method was used to estimate the median TtR and its 95% CI for subjects in the ITT population (50% of subjects were expected to have a CR or PR at this time).
Time Frame: 12 months
Population: The ITT population is all treated subjects having at least one baseline and at least one post baseline assessment of the primary efficacy parameter
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intention-to-treat (ITT) Population
Number analyzed (Participants) | 49
months | NA [NA to NA] — The results could not be determined as too few subjects recorded a response event during the 12 month study duration.

5. Secondary Outcome: Duration of Response (DoR) Within 12 Months
Description: The DoR is an estimation of the time from first documented objective response (CR or PR) to the first date of progressive disease (PD) or death due to disease progression for subjects who experienced an objective response within the first 12 months of treatment (combination and maintenance phases).
  The Kaplan-Meier method was used to estimate the median DoR and its 95% CI for subjects in the ITT population who had an objective response.
Time Frame: 12 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intention-to-treat (ITT) Population
Number analyzed (Participants) | 6
months | NA [NA to NA] — The results could not be determined as too few subjects recorded a response event during the 12 month study duration.

6. Secondary Outcome: The Number of Subjects With a Biochemical Response Using Chromogranin-A (CgA) Levels After 6 Months
Description: Blood samples for CgA blood tumour marker analysis were taken at baseline, weeks 12, 24 and at early withdrawal. The biochemical response after 6 months combination treatment was estimated for subjects with abnormal CgA levels at baseline. Abnormal CgA levels were defined as above the upper limit of normal range (≥100 micrograms/litre [mcg/L]).
  Biochemical response based on CgA levels was categorised as: PR (decrease of CgA ≥ 50%, compared to the baseline CgA), SD (decrease < 50 % or an increase ≤25%, compared to the baseline CgA) or PD (defined as an increase ≥25 %, compared to the baseline CgA).
  The number of subjects in each response category at each time point in the combination phase is presented. Analysis was only carried out on subjects in the ITT population who had abnormal CgA at baseline.
Time Frame: 6 months
Population: Subjects in the ITT population with abnormal CgA levels at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Phase
Number analyzed (Participants) | 34
Participants
  Week 12- PD | 8
  Week 12 - SD | 15
  Week 12- PR | 10
  Week 12 - Missing | 1
  Week 24 - PD | 5
  Week 24 - SD | 9
  Week 24 - PR | 7
  Week 24 - Missing | 0
  Early Withdrawal - PD | 1
  Early Withdrawal - SD | 2
  Early Withdrawal - PR | 1
  Early Withdrawal - Missing | 14

7. Secondary Outcome: The Number of Subjects With a Biochemical Response Using CgA Levels After 12 Months
Description: Blood samples for CgA blood tumour marker analysis were taken at baseline, weeks 12, 24, 36, 48 (end of study) and at early withdrawal. The biochemical response after 12 months combination and maintenance treatment was estimated for subjects with abnormal CgA levels at baseline. Abnormal CgA levels were defined as above the upper limit of normal range (≥100 mcg/L).
  Biochemical response based on CgA levels was categorised as: PR (decrease of CgA ≥50 % compared to the baseline CgA), SD (decrease < 50% or an increase ≤ 25% compared to the baseline CgA) or PD (defined as an increase ≥ 25%, compared to the baseline CgA).
  The number of subjects in each response category at each time point in the maintenance phase is presented. Analysis was only carried out on subjects in the ITT population who had abnormal CgA at baseline.
Time Frame: 12 months
Population: Subjects in the ITT population with abnormal CgA levels at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase - Functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, No Treatment
Number analyzed (Participants) | 5 | 9 | 9
Participants
  Week 24 - PD | 2 | 1 | 2
  Week 24 - SD | 3 | 4 | 2
  Week 24 - PR | 0 | 3 | 3
  Week 24 - Missing | 0 | 1 | 2
  Week 36 - PD | 1 | 1 | 3
  Week 36 - SD | 2 | 4 | 2
  Week 36 - PR | 0 | 1 | 4
  Week 36 - Missing | 0 | 1 | 0
  Week 48 - PD | 1 | 1 | 2
  Week 48 - SD | 0 | 2 | 3
  Week 48 - PR | 1 | 2 | 1
  Week 48 - Missing | 0 | 0 | 0
  Early Withdrawal - PD | 1 | 2 | 1
  Early Withdrawal - SD | 0 | 0 | 0
  Early Withdrawal - PR | 0 | 1 | 1
  Early Withdrawal - Missing | 2 | 0 | 0

8. Secondary Outcome: The Number of Subjects With a Biochemical Response Using 5-Hydroxy-Indol-Amino-Acid (HIAA) Levels After 6 Months
Description: Urine samples for 5-HIAA urinary tumour marker analysis were taken at at baseline, weeks 12, 24and early withdrawal.
  Biochemical response based on 5-HIAA levels was categorised as: Response (5-HIAA reduction compared to baseline) or Progression (5-HIAA increase compared to baseline).
  The number of subjects in each response category at each time point in the combination phase is presented. Analysis was only carried out on subjects in the ITT population with functioning NET.
Time Frame: 6 months
Population: Subjects in the ITT population with functioning NET.
Measure: Count of Participants; unit: Participants
Groups:
- Combination Phase - Functioning NET: All subjects in the combination phase who were categorised at baseline as having functioning NET.
Arm/Group | Combination Phase - Functioning NET
Number analyzed (Participants) | 17
Participants
  Week 12 - Progression | 4
  Week 12 - Response | 6
  Week 12 - Not evaluable | 1
  Week 12 - Missing | 6
  Week 24 - Progression | 6
  Week 24 - Response | 3
  Week 24 - Not evaluable | 1
  Week 24 - Missing | 3
  Early Withdrawal - Progression | 0
  Early Withdrawal - Response | 1
  Early Withdrawal - Not Evaluable | 0
  Early Withdrawal - Missing | 7

9. Secondary Outcome: The Number of Subjects With a Biochemical Response Using 5-HIAA Levels After 12 Months
Description: Urine samples for 5-HIAA urinary tumour marker analysis were taken at baseline, weeks 12, 24, 36, 48 (end of study) and early withdrawal.
  Biochemical response based on 5-HIAA levels was categorised as: Response (5-HIAA reduction compared to baseline) or Progression (5-HIAA increase compared to baseline).
  The number of subjects in each response category at each time point in the maintenance phase is presented. Analysis was only carried out on subjects in the ITT population with functioning NET.
Time Frame: 12 months
Population: Subjects in the ITT population with functioning NET.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase - Functioning NET, Lanreotide
Number analyzed (Participants) | 11
Participants
  Week 24 - Progression | 6
  Week 24 - Response | 3
  Week 24 - Not evaluable | 1
  Week 24 - Missing | 1
  Week 36 - Progression | 3
  Week 36 - Response | 3
  Week 36 - Not evaluable | 0
  Week 36 - Missing | 3
  Week 48 - Progression | 4
  Week 48 - Response | 2
  Week 48 - Not evaluable | 0
  Week 48 - Missing | 2
  Early Withdrawal - Progression | 0
  Early Withdrawal - Response | 0
  Early Withdrawal - Not evaluable | 0
  Early Withdrawal - Missing | 3

10. Secondary Outcome: The Number of Subjects With a Symptomatic Response After 6 Months
Description: Symptomatic response was evaluated as absolute change from baseline in the number of episodes of the lead symptoms (i.e. diarrhoea and flushing) using the mean of the last 3 days before the visit, at each visit, as compared to baseline.
  Symptomatic responses were categorised as: Reduction, Increase or Stability of occurrences of diarrhoea / Reduction, Increase or Stability of occurrences of flushing.
  The number of subjects in each response category at week 24 (end of the combination phase) is presented. Analysis was only carried out on subjects in the ITT population with functioning NET.
Time Frame: 6 months
Population: Subjects in the ITT population with functioning NET.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Phase - Functioning NET
Number analyzed (Participants) | 17
Participants
  Diarrhoea - Reduction | 4
  Diarrhoea - Increase | 2
  Diarrhoea - Stability | 5
  Diarrhoea - Missing | 6
  Flushing - Reduction | 4
  Flushing - Increase | 4
  Flushing - Stability | 3
  Flushing - Missing | 6

11. Secondary Outcome: The Number of Subjects With a Symptomatic Response After 12 Months - Maintenance Phase
Description: Symptomatic response was evaluated as absolute change from baseline in the number of episodes of the lead symptoms (i.e. diarrhoea and flushing) using the mean of the last 3 days before the visit, at each visit, as compared to baseline.
  Symptomatic responses were categorised as: Reduction, Increase or Stability of occurrences of diarrhoea / Reduction, Increase or Stability of occurrences of flushing.
  The number of subjects in each response category at week 48 (end of study) is presented. Analysis was only carried out on subjects in the ITT population with functioning NET.
Time Frame: 12 months
Population: Subjects in the ITT population with functioning NET.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase - Functioning NET, Lanreotide
Number analyzed (Participants) | 11
Participants
  Diarrhoea - Reduction | 4
  Diarrhoea - Increase | 1
  Diarrhoea - Stability | 3
  Diarrhoea - Missing | 3
  Flushing - Reduction | 2
  Flushing - Increase | 3
  Flushing - Stability | 3
  Flushing - Missing | 3

12. Secondary Outcome: European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life (QoL) Core 30 Questionnaire (QLQ-C30): Mean Change From Baseline at 6 Months
Description: Subjects were instructed to complete the QLQ-C30 questionnaire at baseline, weeks 12, 24 or at early withdrawal. The first 28 questions used a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) for evaluating 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (fatigue, nausea/vomiting, pain) & 6 other single items. The last 2 questions represented subject's assessment of overall health & quality of life, coded on a 7-point scale (1=very poor to 7=excellent). The mean change from baseline at week 24 (end of the combination phase) is presented for global health status (scoring of questions 29 & 30) and 5 functional scales, 3 symptom scales and other single items (scoring of questions 1 to 28). Each individual subscore was transformed to range from 0 to 100. A higher score represents a higher level response. Thus, a better QoL/a better level of functioning/a worse level of symptoms.
Time Frame: 6 months
Population: Only subjects in the ITT Population with data available at the week 24 time point were analysed. Only subjects with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combination Phase
Number analyzed (Participants) | 34
units on a scale
  Global health status | -4.9 (18.2)
  Physical functioning | -9.6 (19.4)
  Role functioning | -8.3 (27.6)
  Emotional functioning | -4.7 (17.7)
  Cognitive functioning | -5.9 (15.8)
  Social functioning | -11.8 (23.8)
  Fatigue | 6.9 (20.1)
  Nausea and vomiting | 6.9 (14.9)
  Pain | -1.0 (31.0)
  Dyspnoea | 12.7 (30.7)
  Insomnia: number analyzed (Participants) | 32
  Insomnia | 0.0 (34.9)
  Appetite loss | 2.0 (24.5)
  Constipation | 6.9 (33.6)
  Diarrhoea | -3.9 (34.6)
  Financial difficulties | 2.9 (17.1)

13. Secondary Outcome: EORTC QoL Questionnaire QLQ-C30: Mean Change From Baseline at 12 Months
Description: Subjects were instructed to complete QLQ-C30 questionnaire at baseline, weeks 12, 24, 36, 48 (end of study) or at early withdrawal. The first 28 questions used a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) for evaluating 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (fatigue, nausea/vomiting, pain) & 6 other single items. The last 2 questions represented subject's assessment of overall health & quality of life, coded on a 7-point scale (1=very poor to 7=excellent). The mean change from baseline at week 48 (end of study) is presented for global health status (scoring of questions 29 & 30) and 5 functional scales, 3 symptom scales and other single items (scoring of questions 1 to 28). Each individual subscore was transformed to range from 0 to 100. A higher score represents a higher level response. Thus, a better QoL/a better level of functioning/a worse level of symptoms.
Time Frame: 12 months
Population: Only subjects in the ITT Population with data available at the week 48 time point were analysed. Only subjects with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Phase - Functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, No Treatment
Number analyzed (Participants) | 5 | 8 | 7
units on a scale
  Global health status | -11.7 (40.7) | -3.1 (10.9) | -7.1 (15.5)
  Physical functioning | 8.0 (22.8) | -12.5 (17.6) | -11.4 (13.7)
  Role functioning | 3.3 (29.8) | -2.1 (20.8) | -7.1 (13.1)
  Emotional functioning | 15.0 (19.0) | -6.2 (20.3) | -6.0 (12.5)
  Cognitive functioning | 3.3 (24.7) | -2.1 (20.8) | 2.4 (6.3)
  Social functioning | 13.3 (34.2) | -22.9 (34.4) | -4.8 (15.9)
  Fatigue | -22.2 (30.4) | -9.7 (24.1) | 4.8 (16.8)
  Nausea and vomiting | -10.0 (14.9) | 4.2 (23.1) | 2.4 (6.3)
  Pain | -13.3 (32.1) | 4.2 (24.8) | 9.5 (23.3)
  Dyspnoea: number analyzed (Participants) | 4 | 8 | 7
  Dyspnoea | -8.3 (41.9) | 4.2 (33.0) | 9.5 (16.3)
  Insomnia: number analyzed (Participants) | 5 | 8 | 6
  Insomnia | -13.3 (50.6) | -8.3 (34.5) | 16.7 (27.9)
  Appetite loss | 0.0 (23.6) | 0.0 (39.8) | 14.3 (17.8)
  Constipation | 20.0 (38.0) | -4.2 (11.8) | -4.8 (35.6)
  Diarrhoea | -40.0 (36.5) | 8.3 (15.4) | 0.0 (27.2)
  Financial difficulties | 6.7 (14.9) | 4.2 (27.8) | 9.5 (25.2)

14. Secondary Outcome: Quality of Life Gastrointestinal Neuroendocrine Tumour 21 Questionnaire (QLQ-GI.NET21): Mean Change From Baseline at 6 Months
Description: Subjects were instructed to complete the QLQ-GI.NET21 questionnaire at baseline, weeks 12, 24 or at early withdrawal. It contained 21 questions that used a 4-point scale (1 = Not at all, 2 = A little, 3 = Quite a bit, 4 = Very much) to evaluate 3 defined multi-item symptom scales (endocrine, gastrointestinal and treatment related side effects), 2 single item symptoms (bone/muscle pain and concern about weight loss), 2 psychosocial scales (social function and disease-related worries) and 2 other single items (sexuality and communication). Each individual subscore was transformed to range from 0 to 100. The mean change from baseline at week 24 (end of combination phase) is presented with a higher score representing a higher level response. Thus, a better level of functioning/a worse level of symptoms.
Time Frame: 6 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Combination Phase
Number analyzed (Participants) | 34
Units on a scale
  Endocrine symptoms | -1.0 (13.5)
  Gastrointestinal (G.I.) symptoms | 5.7 (14.0)
  Treatment related symptoms: number analyzed (Participants) | 14
  Treatment related symptoms | 3.6 (30.1)
  Social function | 2.3 (25.3)
  Disease related worries | 1.6 (27.1)
  Muscle/bone pain symptoms | 1.0 (37.1)
  Body image | 0.0 (23.2)
  Weight gain: number analyzed (Participants) | 31
  Weight gain | -11.8 (30.5)
  Information/communication function: number analyzed (Participants) | 32
  Information/communication function | -9.4 (22.8)
  Sexual function: number analyzed (Participants) | 14
  Sexual function | -4.8 (17.8)

15. Secondary Outcome: QoL Questionnaire QLQ-GI.NET21: Mean Change From Baseline at 12 Months
Description: Subjects were instructed to complete the QLQ-GI.NET21 questionnaire at baseline, weeks 12, 24, 36, 48 (end of study) or at early withdrawal. It contained 21 questions that used a 4-point scale (1 = Not at all, 2 = A little, 3 = Quite a bit, 4 = Very much) to evaluate 3 defined multi-item symptom scales (endocrine, gastrointestinal and treatment related side effects), 2 single item symptoms (bone/muscle pain and concern about weight loss), 2 psychosocial scales (social function and disease-related worries) and 2 other single items (sexuality and communication). Answers were converted into grading scale, with values between 0 and 100. Each individual subscore was transformed to range from 0 to 100. The mean change from baseline at week 48 (end of study) is presented with a higher score representing a higher level response. Thus, a better level of functioning/a worse level of symptoms.
Time Frame: 12 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Phase - Functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, No Treatment
Number analyzed (Participants) | 5 | 8 | 7
units on a scale
  Endocrine symptoms | -13.3 (21.4) | -5.6 (19.7) | 1.6 (4.2)
  G.I. symptoms | -4.0 (21.9) | 0.0 (19.2) | 6.7 (7.7)
  Treatment related symptoms: number analyzed (Participants) | 2 | 3 | 0
  Treatment related symptoms | 0.0 (0.0) | -11.1 (34.7) |
  Social function | -6.7 (23.0) | 9.7 (20.9) | -6.3 (16.8)
  Disease related worries | -6.7 (36.5) | 1.4 (15.1) | -3.2 (30.6)
  Muscle/bone pain symptoms | -6.7 (14.9) | 4.2 (33.0) | 4.8 (30.0)
  Body image | 0.0 (23.6) | 4.2 (27.8) | 4.8 (12.6)
  Weight gain: number analyzed (Participants) | 5 | 7 | 7
  Weight gain | -20.0 (29.8) | 9.5 (25.2) | -9.5 (56.8)
  Information/communication function | 0.0 (70.7) | 0.0 (17.8) | -4.8 (12.6)
  Sexual function: number analyzed (Participants) | 2 | 4 | 3
  Sexual function | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

16. Secondary Outcome: DCR by O6-methylguanine-DNA Methyl-transferase (MGMT) Expression and Methylation and Somatostatin Receptor (SSTR) Expression After 6 Months
Description: In all subjects whose tumour tissue was available, MGMT expression/methylation and SSTR expression was analysed. After 6 months, the DCR (SD+PR+CR) by MGMT methylation and expression and by SSTR 2a and SSTR 5 expression was evaluated.
  DCR in response to MGMT methylation and expression results are presented. SSTR 2a and SSTR 5 expression is categorised as: No Receptors, Cytoplasmatic Expression (CE), Focal Expression (FE), Complete Circumferent Membrane Expression (CCME).
  The DCR was defined as the proportion of subjects with a response of CR, PR or SD after 6 months of combination treatment within each methylation/expression category. The DCR was described in the ITT population along with its 95% CI and was compared to 45% with an exact binomial proportion test.
Time Frame: 6 months
Population: Percentages are based on the number of subjects in the ITT population and with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Combination Phase
Number analyzed (Participants) | 49
percentage of subjects
  MGMT Methylation: number analyzed (Participants) | 9
  MGMT Methylation | 100.0 [66.4 to 100.0]
  MGMT No methylation: number analyzed (Participants) | 13
  MGMT No methylation | 84.6 [54.6 to 98.1]
  MGMT Expression: number analyzed (Participants) | 11
  MGMT Expression | 90.9 [58.7 to 99.8]
  MGMT No expression: number analyzed (Participants) | 20
  MGMT No expression | 70.0 [45.7 to 88.1]
  SSTR 2a No Receptors: number analyzed (Participants) | 0
  SSTR 2a CE: number analyzed (Participants) | 0
  SSTR 2a FE: number analyzed (Participants) | 15
  SSTR 2a FE | 86.7 [59.5 to 98.3]
  SSTR 2a CCME: number analyzed (Participants) | 22
  SSTR 2a CCME | 72.7 [49.8 to 89.3]
  SSTR 5 - No Receptors: number analyzed (Participants) | 24
  SSTR 5 - No Receptors | 75.0 [53.3 to 90.2]
  SSTR 5 CE: number analyzed (Participants) | 2
  SSTR 5 CE | 100.0 [15.8 to 100.0]
  SSTR 5 FE: number analyzed (Participants) | 11
  SSTR 5 FE | 81.8 [48.2 to 97.7]
  SSTR 5 CCME: number analyzed (Participants) | 0

17. Secondary Outcome: Pharmacokinetic (PK) Results: Lanreotide ATG 120 mg Serum Concentrations Within 12 Months
Description: Lanreotide ATG levels were measured in a subset of subjects to evaluate if temozolomide co-treatment had an impact on lanreotide serum concentration over a 12 month period.
  Blood samples were collected for the determination of lanreotide ATG in serum at baseline, weeks 4, 12, 24 and 48 (end of study).
  The concentrations of lanreotide ATG in serum were determined by a validated radioimmunoassay analysis method with a lower limit of quantitation of 0.08 nanograms [ng]/mL).
  Serum concentrations of lanreotide ATG at each of the time points in the combination and maintenance phase are presented. Only subjects with data available for analysis are presented.
Time Frame: Baseline (week 1) and weeks 4, 12, 24 and 48
Population: PK analysis was performed using the valid PK population.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PK Subset: All subjects for whom PK assessments were performed and with evaluable PK data.
Arm/Group | PK Subset
Number analyzed (Participants) | 16
ng/mL
  Baseline | 0.44 (1.22)
  Week 4: number analyzed (Participants) | 14
  Week 4 | 2.45 (1.16)
  Week 12: number analyzed (Participants) | 11
  Week 12 | 5.06 (3.01)
  Week 24: number analyzed (Participants) | 9
  Week 24 | 5.83 (1.93)
  Week 48: number analyzed (Participants) | 7
  Week 48 | 3.68 (3.36)

ADVERSE EVENTS:
Time Frame: 13 months (12 month study treatment plus 28 days)
Description: Treatment Emergent Adverse Events (TEAEs) are reported for both the combination and maintenance phases and include events with an onset after the start of study drug treatment to the last intake of study drug plus 28 days.
Groups:
- Maintenance Phase - Functioning NET, Lanreotide: In case of clinical benefit, defined as either CR, PR or SD, after the first 6 months combination phase all subjects with functioning NET continued to receive lanreotide ATG 120 mg for another 6 months. This maintenance phase started with visit 8, week 24.
Arm/Group | Combination Phase | Maintenance Phase - Functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, Lanreotide | Maintenance Phase - Non-functioning NET, No Treatment
All-Cause Mortality (participants affected / at risk) | 1/57 | 1/11 | 1/14 | 1/12
Serious Adverse Events (participants affected / at risk) | 17/57 | 3/11 | 4/14 | 4/12
Other Adverse Events (participants affected / at risk) | 52/57 | 9/11 | 13/14 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Phase (N=57) | Maintenance Phase - Functioning NET, Lanreotide (N=11) | Maintenance Phase - Non-functioning NET, Lanreotide (N=14) | Maintenance Phase - Non-functioning NET, No Treatment (N=12)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular vascular disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Phase (N=57) | Maintenance Phase - Functioning NET, Lanreotide (N=11) | Maintenance Phase - Non-functioning NET, Lanreotide (N=14) | Maintenance Phase - Non-functioning NET, No Treatment (N=12)
Anaemia (Blood and lymphatic system disorders) | 7 (9) | 0 (0) | 0 (0) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 6 (8) | 0 (0) | 0 (0) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 8 (10) | 0 (0) | 2 (2) | 4 (8)
Neutropenia (Blood and lymphatic system disorders) | 6 (7) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (28) | 1 (1) | 3 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (6) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ocular vascular disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (7) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 12 (22) | 2 (3) | 4 (6) | 2 (2)
Anal inflammation (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (16) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 21 (35) | 0 (0) | 3 (4) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 10 (16) | 1 (1) | 2 (3) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 24 (55) | 1 (1) | 4 (5) | 1 (1)
Pancreatic insufficiency (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Steatorrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 19 (40) | 1 (1) | 2 (3) | 1 (1)
Administration site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 19 (32) | 2 (2) | 4 (4) | 5 (7)
Feeling cold (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 1 (1) | 3 (4) | 3 (8)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (8) | 3 (4) | 2 (3) | 3 (3)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 6 (6) | 1 (2) | 1 (1) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 8 (8) | 0 (0) | 2 (2) | 3 (3)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (9) | 1 (1) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (6) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 7 (9) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 3 (5) | 1 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 1 (1) | 2 (2) | 2 (2)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication of the Study Results shall be made without the Sponsor's prior written approval which shall not be unreasonably withheld. Sponsor must be provided with the final version of any abstract, presentation or paper before submission, and the Sponsor shall provide scientific comments within 2 weeks for an abstract or presentation or 6 weeks for an article. If no comments are received within these periods, this silence of Sponsor can be considered as approval to proceed to publication.